CLINICAL TRIAL: NCT00717600
Title: Bacteriuria Eradication Through Probiotics
Acronym: BERP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Baylor College of Medicine (Other)
Collaborators: Chr Hansen (Industry); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Eric A. Jones, Texas Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-21679
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2008-07-17 (Estimated); Status verified 2008-07

CONDITIONS: Bacteriuria
Keywords: bacteriuria; urinary tract infection; probiotics; lactobacillus; vagina; bladder; neurogenic bladder; spina bifida; myelomeningocele; neuropathic bladder
MeSH Terms: conditions — Bacteriuria; Urinary Tract Infections; Urinary Bladder, Neurogenic; Spinal Dysraphism; Meningomyelocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Oral probiotics
  Interventions: Dietary Supplement: Lactobacillus reuteri RC-14 and Lactobacillus rhamnosus GR-1

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri RC-14 and Lactobacillus rhamnosus GR-1 — 2x10^9 cfu of Lactobacillus reuteri RC-14 and Lactobacillus rhamnosus GR-1 administered daily via a single orally ingested freeze-dried capsule.
  Other Names: Lactobacillus reuteri RC-14 and Lactobacillus rhamnosus GR-1 (Urex cap-5 from CHR. Hansen), batch 2750558

SUMMARY:
Many children who catheterize their bladders because of spina bifida or other neurologic disorders have bacteriuria. This can lead to urinary tract infections by bacteria from the gut which colonize the vagina and are carried into the bladder during catheter passage. We seek to test whether oral administration of probiotic bacteria can "displace" these vagina-derived uropathogens and reduce or prevent bacteriuria in girls with spina bifida who empty their bladders through catheterization.

DETAILED DESCRIPTION:
In children with spina bifida and neurogenic bladder dysfunction, the need for intermittent bladder catheterization increases the risk of bacteriuria. In many patients, this leads to a clinically significant urinary tract infection (UTI). Many of these children are placed on long term, low dose antibiotic suppression to prevent recurrent urinary infection. Unfortunately, bacteriuria often persists despite daily antibiotic therapy, and breakthrough urinary tract infections are common. Furthermore, this approach carries the potential for deleterious side effects, and may promote the development of antibiotic-resistant bacteria.

Urinary tract infection in girls occurs when virulent bacteria migrate from the rectum and colonize the vagina and peri-urethral mucosa, thus gaining access to the bladder. In girls with spina bifida, access to the bladder is greatly facilitated by catheter passage. Antibiotic prophylaxis relies on maintaining a low dose of antibiotic in the urinary stream, which decreases peri-urethral colonization, and prevents proliferation of bacteria after they gain access to the bladder. An alternative approach to daily antibiotic prophylaxis is to decrease the risk of urinary colonization with virulent bacteria by supplementing the normal bacteria flora with non-infection causing strains of bacteria.

Probiotics are dietary supplements containing potentially beneficial bacterial strains such as Lactobacillus. The safety of oral administration of probiotics has been demonstrated in several studies over the last 30 years. Studies using L. rhamnosus GG, a probiotic introduced in the late 1980s to alleviate diarrhea, have shown promising results when used for UTI prevention. In one study, researchers found that the subjects consuming Lactobacillus GG drinks had fewer episodes of UTI compared to those women not receiving probiotics. A placebo-controlled study in premature infants also used L. rhamnosus GG in an attempt to prevent UTI. The number of urinary infections was reduced but statistically the difference was not significant. Finally, a recent randomized clinical trial demonstrated that the rate of UTI in patients taking prophylactic antibiotics was similar to that of patients taking Lactobacillus acidophilus alone. The efficacy of probiotic usage in the spina bifida population has not been reported.

Our objective is to determine whether over the course of 3 months, probiotics can reduce preexisting or new bacteriuria in girls with spina bifida who perform clean intermittent catheterization for bladder emptying. We will also attempt to ascertain whether changes in bacteriuria are associated with vaginal colonization by the administered probiotics.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects are girls (age 3 months to 18 years) with spina bifida as a sole urologic diagnosis
* perform clean intermittent catheterization because of neurogenic bladder.
* Secondary vesicoureteral reflux is permissible.
* Patients with appendicovesicostomies and no other forms of urinary diversion are permitted.

Exclusion Criteria:

* Patients will be excluded if they are taking antibiotics
* immunosuppressed, i.e., transplant recipients or children with congenital immunodeficiencies
* poorly controlled diabetes
* untreated HIV infection
* immunosuppression from corticosteroids
* malnutrition
* pregnancy
* chronic indwelling catheters in the bladder
* any urinary diversion or bladder augmentation.

Max Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-09 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
bacteriuria | 3 months

SECONDARY OUTCOMES:
urinary tract infections | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Jones, M.D., Principal Investigator — Texas Children's Hospital, Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States